CLINICAL TRIAL: NCT03684083
Title: Inflammatory Response to Paramyxovirus Infection in an Ex-vivo Model of Bronchial Epithelial Cells in Allogeneic Hematopoietic Stem Cell Recipients
Brief Title: Inflammatory Response to Paramyxovirus Infection in an Ex-vivo Model of Bronchial Epithelial Cells in Allogeneic HSCT Recipients
Acronym: ALLOVIRO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01325-48
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pulmonary biopsy with transcriptomic analysis after cell infection by parainfluenza virus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: patients having received heterologous stem cell transplantation (HSCT)
  Interventions: Procedure: bronchial biopsies
- Control: patients without HSCT
  Interventions: Procedure: bronchial biopsies

INTERVENTIONS:
Procedure: bronchial biopsies — bronchial fibroscopy with bronchial biopsies

SUMMARY:
Introduction. Chronic graft-versus-host-disease (GVHD) is the main late noninfectious complication after allogeneic hematopoietic stem cell transplantation (HSCT) that can affect several organs. Bronchiolitis obliterans syndrome (BOS) is recognized as pulmonary chronic GVHD. A diagnosis of a lower respiratory tract infection in the first 100 days following transplant has been associated to the development of BOS. One hypothesis is that the first stage driving to BOS is a previous aggression of bronchial epithelial cells by various factors such as chemotherapy and radiotherapy. Thereafter, data suggest that viral infections, in particular Parainfluenza viruses could be a trigger for BOS. The alloimmune reaction activated by the respiratory virus could lead to the fibrosis process. Our hypothesis is that the bronchial epithelium of allogeneic HSCT recipients has phenotypic specificities that are associated with a specific response to the viral respiratory infections (in particular paramyxovirus) leading to the development of BOS.

Main objective. To characterize and compare the inflammatory response after infection with Parainfluenza 3 virus in an ex-vivo model of bronchial epithelial cells obtained from allogeneic HSCT recipients and controls.

Objective secondary. To characterize the phenotypic specificities of allogeneic HSCT recipients' bronchial epithelium.

Methodology, and experimental plan. Prospective, monocentric research. Bronchial biopsies obtained from patients, will be completely differentiated after 21 days of culture. Epithelial cells will be infected by the virus strain Parainfluenza 3. Transcriptome of the cells from both allogeneic HSCT patients and controls, infected and non-infected will be analyzed 48 hours after infection.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT patients [case]
* requirement of ng bronchial fibroscopy with bronchial biopsies for the exploration of FEV1 decline [case]
* non Allogeneic HSCT patients [control]
* .requirement of bronchial fibroscopy for exploration of a lung mass or of interstitial lung disease, requiring bronchial biopsies [control]

Exclusion Criteria:

* Minor or major patients protected
* Radiotherapy or chemotherapy [control group]
* Respiratory infection
* History of smoking >= 15 packs/yr

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case study population: patients having received Allogeneic HSCT Control study population : patients without Allogeneic HSCT
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cells Transcriptome after infection by parainfluenza virus | 21 days
  inflammatory response after infection with Parainfluenza 3 virus in an ex-vivo model of bronchial epithelial cells assessed by cells transcriptome

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Hospital, Paris, France